CLINICAL TRIAL: NCT03600610
Title: Evaluation of CARdiac Morphological and Functional Abnormalities by Echocardiography and Magnetic Resonance Imaging in Malnourished Patients Suffering From Anorexia Nervosa
Brief Title: Evaluation of CARdiac Abnormalities by Echocardiography and MRI in Malnourished Patients Suffering From Anorexia Nervosa
Acronym: CARERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-22
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Anorexia Nervosa; Cardiac Anomaly
MeSH Terms: conditions — Anorexia Nervosa; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group (Experimental): malnourished patients with anorexia nervosa gadolinium-enhanced cardiac MRI will be performed
  Interventions: Device: gadolinium-enhanced cardiac MRI
- control group (Active Comparator): age- and sex- matched, normal weight, healthy volunteers gadolinium-enhanced cardiac MRI will be performed
  Interventions: Device: gadolinium-enhanced cardiac MRI

INTERVENTIONS:
Device: gadolinium-enhanced cardiac MRI — cardiac magnetic resonance imaging with gadolinium injection used T1-Mapping

SUMMARY:
Anorexia nervosa is an eating disorder occurring in adolescent females, characterized by voluntary dietary restriction, intense fear of gaining weight, and disturbed body image perception. Anorexia nervosa is characterized by the potential severity of its prognosis. While complete remission occurs in about 50% of cases, up to 20% of patients will develop a chronic relapsing form that leads to social disintegration. Moreover, anorexia nervosa has the highest mortality rate among psychiatric diseases with a risk of death of up to 10%. 30% of deaths in anorexia nervosa are attributed to cardiac complications remaining insufficiently described, and their screening at a preclinical stage is still poorly codified. Echocardiography findings show reduced left ventricular mass, pericardial effusion or mitral valve prolapse ; in addition, systolic function appears to be preserved whereas a global diastolic dysfunction, estimated with trans-mitral flow and global longitudinal strain. While the interest of cardiac echography has been well established, only one study used MRI as a means of cardiac evaluation in anorexia nervosa: interestingly, local myocardial fibrosis is pointed and could potentially contribute to cardiac rhythm disorders. No study has yet used T1-Mapping MRI to evaluate if diffuse myocardial fibrosis is prevalent in this population group.

The investigators conduct a transversal, observational, monocentric study whereby malnourished patients with anorexia nervosa and age- and sex- matched, normal weight, healthy volunteers will undergo a gadolinium-enhanced cardiac MRI. The primary objective of this study is to evaluate and compare the frequency of cardiac fibrosis in those populations. Other cardiac MRI parameters will be described and compared as secondary objectives. Moreover, non-cardiac parameters evaluated by MRI such as adipose tissue distribution in anorexia nervosa patients compared with controls.

In addition, patients with anorexia nervosa, a clinical, morphological and biological evaluation, including anthropometric parameters, biphotonic absorptiometry, resting electrocardiogram, cardiac echography and classical biological markers of malnutrition, will be done.

DETAILED DESCRIPTION:
Anorexia nervosa is an eating disorder occurring most frequently in adolescent females, characterized by 1/ voluntary dietary restriction, leading to lower than normal body weight and, often, loss of considerable amount of weight and, thereby, malnutrition, 2/ intense fear of gaining weight, even when the individual is already underweight, starved or malnourished and 3/ disturbed body image perception, including extreme emphasis on the appearance. Anorexia nervosa is characterized by the potential severity of its prognosis. While complete remission occurs in about 50% of cases, up to 20% of patients will develop a chronic relapsing form that leads to social disintegration. Moreover, anorexia nervosa has the highest mortality rate among psychiatric diseases with a risk of death of up to 10% (including suicide and clinical complications of severe malnutrition). If approximatively 30% of deaths in anorexia nervosa are attributed to cardiac complications, the nature and the frequency of such complications remain insufficiently described, and their screening at a preclinical stage is still poorly codified. Echocardiography findings are well documented and include reduced left ventricular mass, pericardial effusion (in 22 to 35% of cases), or mitral valve prolapse (in up to 35% of cases); in addition, systolic function, evaluated by the ejection fraction appears to be preserved whereas a global diastolic dysfunction, estimated with trans-mitral flow and global longitudinal strain, is reported. While the interest of cardiac echography has been well established, only one study used MRI (magnetic resonance imaging) as a means of cardiac evaluation in anorexia nervosa: interestingly, this study found local myocardial fibrosis in nearly 25% of patients with anorexia nervosa, which could potentially contribute to cardiac rhythm disorders. That said, no study has yet used T1-Mapping MRI to evaluate if diffuse myocardial fibrosis is prevalent in this population group.

The investigators aim to conduct a transversal, observational, monocentric study whereby malnourished patients with anorexia nervosa (n = 38) and age- and sex- matched, normal weight, healthy volunteers (n = 38) will undergo a gadolinium-enhanced cardiac MRI. The primary objective of this study is to evaluate and compare the frequency of cardiac fibrosis in those populations using cardiac MRI. Other morphological and functional cardiac MRI parameters will be described and compared as secondary objectives: local myocardial fibrosis using enhanced MRI; myocardial and left ventricular mass; myocardial triglyceride quantification using Proton spectroscopy; cardiac high-energy metabolism using Phosphore-31 spectroscopy. Moreover, non-cardiac parameters evaluated by MRI such as adipose tissue distribution (visceral fat, liver fat, bone marrow fat) in anorexia nervosa patients compared with controls.

In addition, patients with anorexia nervosa, a clinical, morphological and biological evaluation, including anthropometric parameters, biphotonic absorptiometry, resting electrocardiogram, cardiac echography and classical biological markers of malnutrition, will be done. Multivariate analysis will then be used to identify possible correlating factors between cardiac MRI findings and clinical, morphological and biological parameters in malnourished patients with anorexia nervosa, so as to shed light on possible new risk stratification models or predictive tools for cardiac complications that could be later evaluated by appropriate studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Anorexia nervosa as defined by DSM-V with BMI < 15kg/m²
* Healthy controls with BMI within 18 to 25 kg/m²

Exclusion Criteria:

* History of cardiac disease previous to the diagnosis of anorexia nervosa
* On-going pregnancy or previous 3 month
* Breast feeding
* RMI contraindication
* History of allergic reaction to contrast product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Diffuse myocardial fibrosis | 45 minutes
  Cardiac MRI (T1 Mapping shMOLLI) Diffuse myocardial fibrosis will be measured using ShMOLLI type T1 mapping methods to obtain high-resolution maps in the heart and a quantitative measure of fibrosis

SECONDARY OUTCOMES:
Local myocardial fibrosis | 45 minutes
  Cardiac MRI (Late Gadolinium enhancement) Nodular myocardial fibrosis will be measured using late gadolinium enhancement after DOTAREM-gadolinium single dose injection (0.1 mmol / kg)
Myocardial triglycerides quantification | 1hour
  quantification by Proton spectroscopy A T1 contrast sequence is used with a set of small-axis sections (n = 14) covering the entire heart for evaluation of pericardial adipose tissue volume
Cardiac metabolism | 1day
  Phosphore-31 spectroscopy It will be evaluated by spectroscopy of phosphorus 31 (SRM-P31) with the study of phosphocreatine / adenosine triphosphate ratio

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Pubique Des Hopitaux de Marseille, Marseille, PACA, France